CLINICAL TRIAL: NCT02657668
Title: Pilot Study of Efficacy of Emotion Focused Therapy on Stress, Resiliency and Coping Strategies in Irritable Bowel Syndrome Patients
Brief Title: Emotion Focused Therapy in Irritable Bowel Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Islamic Azad University, Najafabad Branch (Other)
Responsible Party: Principal Investigator, Sayed Abbas Haghayegh, Assisstant professor, Islamic Azad University, Najafabad Branch
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IslamicAUN
Record Dates: First submitted 2016-01-07; First posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Irritable Bowel Syndrome; Emotion Focused Therapy; Stress; Resilience; Coping Strategies
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome | interventions — Emotion-Focused Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): Emotion focused therapy: EFT was conducted in eight sessions (without pretest and posttest sessions) according to Greenberg's manual (22) in a clinic of gastrointestinal patients. According to Greenberg manual, EFT consists of three steps: 1) emotional awareness 2) accessing healthy emotions 3) skills of emotional intelligence. There were five individuals in the posttest (because of being absent more than three sessions or not participating in the posttest).
  Interventions: Behavioral: Emotion Focused Therapy
- Control Group (No Intervention): Control group: For control group interactions to be effective in therapeutic outcomes, the psycho-educational group was assigned as control group. The Psycho-educational group was conducted in four sessions (without pretest and posttest sessions). They became familiar with etiology and role of psychological factors in IBS, without any psychotherapy. Eight members were removed (because of being absent more than three sessions).

INTERVENTIONS:
Behavioral: Emotion Focused Therapy — EFT was conducted in eight sessions (without pretest and posttest sessions) according to Greenberg's manual (22) in a clinic of gastrointestinal patients. According to Greenberg manual, EFT consists of three steps: 1) emotional awareness 2) accessing healthy emotions 3) skills of emotional intelligence. There were five individuals in the posttest (because of being absent more than three sessions or not participating in the posttest).
  Other Names: EFT
  Arms: Treatment Group

SUMMARY:
The study was quasi-experimental including patients in two intervention and control groups. Three measurements were done: pretest, post-test, and a two-months follow-up. The study population included patients with irritable bowel syndrome(diagnosed by specialists and based on the criteria of Rome III), who referred to a general Hospital. Fifty two irritable bowel syndrome patients were selected and assigned to two experiment (26 cases) and control (26 cases) groups. The criteria below were considered in selection of patients.

Inclusion criteria: 1) Patients should not have participated in other psychological interventions concurrently; 2) Participants had not reported diagnosis of non-functional gastrointestinal illnesses. 3) Women patients had not been in pregnancy; 4) Participants had not met diagnosis of schizophrenia and bipolar disorders.

Exclusion criteria: Three or more absences in the group sessions Co-variate variables: 1) demo-graphical variables (age, birth order, and education); 2) clinical variables (global psychological status, mind-body attribution, and duration of disease).

DETAILED DESCRIPTION:
The study was quasi-experimental including patients in two intervention and control groups. Three measurements were done: pretest, post-test, and a two-months follow-up. The study population included patients with irritable bowel syndrome(diagnosed by specialists and based on the criteria of Rome III), who referred to general Hospital . Fifty two irritable bowel syndrome patients were selected and assigned to two experiment (26 cases) and control (26 cases) groups. The criteria below were considered in selection of patients.

Intervention design Experimental group: Emotion focused therapy was conducted in eight sessions (without pretest and post-test sessions) according to Greenberg's manual (22) in a clinic of gastrointestinal patients. According to Greenberg manual, emotion focused therapy consists of three steps:1) emotional awareness 2) accessing healthy emotions 3) skills of emotional intelligence.There were five individuals in the post-test (because of being absent more than three sessions or not participating in the post-test).

Control group: For control group interactions to be effective in therapeutic outcomes, the psycho-educational group was assigned as control group. The Psycho-educational group was conducted in four sessions (without pretest and post-test sessions). They became familiar with etiology and role of psychological factors in irritable bowel syndrome, without any psychotherapy. Eight members were removed (because of being absent more than three sessions).

Ethical permission This study was approved by the research committee of University of Isfahan. To appreciate participants, after group therapy, the results of therapy were reported to the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should not have participated in other psychological interventions concurrently;
2. Participants had not reported diagnosis of non-functional gastrointestinal illnesses.
3. Women patients had not been in pregnancy;
4. Participants had not met diagnosis of schizophrenia and bipolar disorders.

Exclusion Criteria:

Three or more absences in the group sessions

Covariate variables:

1. demographical variables (age, birth order, and education);
2. clinical variables (global psychological status, mind-body attribution, and duration of disease).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Stress | pretest- post test-follow-up(in 4 month)
  Depression-Anxiety-Stress scale(DASS):DASS was published by Lovibond & Lovibond in 1995.Short form of DASS conclude 21 sentences that each 7 sentences in related to one subscale. In this research, has been used of subscale of stress. Iranian form of this subscale has been significant relation(concurrent validity) with Holms-Rahe stress questionnaire(r:0/49)

SECONDARY OUTCOMES:
Coping Strategies | pretest- post test-follow-up(in 4 month)
  Coping Strategies Questionnaire: This questionnaire was published by Andler and Parker in 1990.This instrument conclude 3 subscales: problem-oriented ,Emotion-oriented strategies and Aversion-oriented strategies. This questionnaire consist 48 questions that are completed in a likert range(1-5).Retest reliability of these subscales has been 0/6,0/61 and 0/64.Internal reliability has been reported higher than 0/7

OTHER OUTCOMES:
Resiliency | pretest- post test-follow-up(in 4 month)
  Resiliency Questionnaire: This questionnaire was published by Connor& Davidson in 2003.This instrument consists 25 questions that are completed in a likert range(0-4).In Iranian form, Internal reliability has been reported 0/89 and construct of this questionnaire has been confirmed in factor analysis

IPD SHARING:
Plan to Share IPD: Yes
according to inclusion and exclusion criteria selected